CLINICAL TRIAL: NCT01452802
Title: Risk Assessment and Comparative Effectiveness of Left Ventricular Assist Device and Medical Management in Ambulatory Heart Failure Patients
Brief Title: Risk Assessment and Comparative Effectiveness of Left Ventricular Assist Device (LVAD) and Medical Management
Acronym: ROADMAP
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TC07272011
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: HeartMate II; heart-assist device; medical management; optimal medical management; Heart Failure NYHA Class IIIB/IV; Thoratec Corporation
MeSH Terms: conditions — Heart Failure | interventions — Practice Management, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HM II (HeartMate II LVAD): Subjects who elect to, and receive HM II LVAD therapy at baseline
  Interventions: Device: HM II (HeartMate II LVAD)
- OMM (Optimal Medical Management): Subjects who elect to remain on optimal medical management
  Interventions: Drug: OMM (Optimal Medical Management)

INTERVENTIONS:
Device: HM II (HeartMate II LVAD) — The HM II pump contains a single moving component, the rotor. The pump is implanted just below the left hemidiaphragm with the inflow attached to the apex of the left ventricle and the outflow graft anastomosed to the ascending aorta. Blood is pumped continuously throughout the cardiac cycle from the left ventricle to the aorta.
  Other Names: Left Ventricular Assist Device
  Groups: HM II (HeartMate II LVAD)
Drug: OMM (Optimal Medical Management) — Optimal medical management per established heart failure guidelines for this subject population including ACE inhibitors, beta blockers and aldosterone antagonists 45 out of the last 60 days or an inability to tolerate neurohormonal antagonists.
  Other Names: Medical Management
  Groups: OMM (Optimal Medical Management)

SUMMARY:
The purpose of this study is to evaluate and compare the effectiveness of the HeartMate II (HM II) Left Ventricular Assist Device (LVAD) support versus OMM in ambulatory NYHA Class IIIB/IV heart failure patients who are not dependent on intravenous inotropic support and who meet the FDA approved indications for HM II LVAD destination therapy.

DETAILED DESCRIPTION:
The HeartMate II (HM II) LVAD is approved by the U.S. Food and Drug Administration (FDA) for use in destination therapy (DT) patients with New York Heart Association (NYHA) Class IIIB/IV symptoms.

The ROADMAP trial is a prospective, multi-center, non-randomized, controlled, observational study that is designed to evaluate the effectiveness of HM II LVAD support versus optimal medical management (OMM) in ambulatory NYHA Class IIIB/IV heart failure patients who are not dependent on intravenous inotropic support and who meet the FDA approved indications for HM II LVAD destination therapy. Subjects will be enrolled in one of two cohorts: OMM or LVAD. Together with the investigator, the subjects will decide which cohort to enter into at their baseline visit. This study will include experienced HM II LVAD implant centers as well as community centers that care for a large volume of heart failure patients. Study patients will be followed for up to 24 months post enrollment for survival, quality of life and functional status.

ELIGIBILITY:
The following are general criteria; more specific criteria are included in the study protocol:

Inclusion Criteria:

* NYHA Class IIIB/IV (refer to Appendix IV for definitions)
* Left ventricular ejection fraction (LVEF) ≤ 25%
* Not currently listed for heart transplantation, and not planned in next 12 months
* On optimal medical management
* Limited functional status as demonstrated by 6MWT <300 meters
* At least:

  * One hospitalization for HF in last 12 months or
  * At least 2 unscheduled emergency room or infusion clinic visits (may include intravenous diuretic therapy, etc.) for HF in last 12 months

Exclusion Criteria:

* Presence of mechanical aortic or mitral valve, including planned conversion to bioprosthesis
* Platelet count < 100,000/mi within 48 prior to enrollment
* Any inotrope use within 30 days prior to enrollment
* Inability to perform 6MWT for any reason
* Any condition, other than heart failure, that could limit survival to less than 2 years
* History of cardiac or other organ transplant
* Existence of any ongoing mechanical circulatory support (including intraaortic balloon pump, temporary circulatory support devices, etc.) at the time of enrollment
* Presence of active, uncontrolled, systemic infection
* History of an unresolved stroke within 90 days prior to enrollment, or a history of cerebral vascular disease with significant (> 80%)extracranial stenosis
* Contraindication to anticoagulation/antiplatelet therapy
* CRT or CRT-D within 3 months prior to enrollment
* Coronary revascularization (e.g. CABG, PCI) within 3 months prior to enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HM II implanting centers and community/referral heart failure clinics
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Composite of survival with improvement in Six Minute Hallway Walk Test distance from baseline of ≥ 75m. | 12 months

SECONDARY OUTCOMES:
Risk stratified subgroup analysis of the primary endpoint and temporal analysis of primary endpoint. | 6, 12, 18, and 24 months
Accuracy of prognostic survival risk models including Seattle Heart Failure Model (SHFM) and HeartMate II Risk Score (HMRS) | Baseline and 6, 12, 18 and 24 months
Actuarial survival and survival free of stroke: a) intent-to-treat; and b) as treated. | 24 months
Survival in LVAD group free of pump replacement. | 24 months
Quality of Life using the EQ-5D-5L Health Utility Index. | Baseline and 6, 12, 18 and 24 months
Depression using Patient Health Questionnaire-9 (PHQ-9). | Baseline and 6, 12, 18 and 24 months
Questionnaire on patient decisions related to LVAD therapy versus optimal medical management. | Baseline and 6, 12, 18 and 24 months
Functional status using 6MWT distance and NYHA Classification | Baseline and 6, 12, 18 and 24 months
Incidence of adverse events, rehospitalizations, days alive and not hospitalized. | 3, 6, 9, 12, 15, 18, 21 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Farrar, PhD, Study Director — Abbott Medical Devices
Locations (52):
- United States (52):
  - Baptist Medical Center, Little Rock, Arkansas
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Keck Medical Center of USC, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Stanford University, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Shands Hospital at University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - St. Joseph's Hospital / Atlanta, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. Vincent's Hospitals and Health Services, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mercer Bucks Cardiology, Robbinsville, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - The Metro Health System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Inc., Oklahoma City, Oklahoma
  - St. John Medical Center, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Milton Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Memorial Hermann, TMC, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - University of Utah Medical School, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Stehlik J, Estep JD, Selzman CH, Rogers JG, Spertus JA, Shah KB, Chuang J, Farrar DJ, Starling RC; ROADMAP Study Investigators. Patient-Reported Health-Related Quality of Life Is a Predictor of Outcomes in Ambulatory Heart Failure Patients Treated With Left Ventricular Assist Device Compared With Medical Management: Results From the ROADMAP Study (Risk Assessment and Comparative Effectiveness of Left Ventricular Assist Device and Medical Management). Circ Heart Fail. 2017 Jun;10(6):e003910. doi: 10.1161/CIRCHEARTFAILURE.116.003910. PMID 28611126
- [Derived] Lanfear DE, Levy WC, Stehlik J, Estep JD, Rogers JG, Shah KB, Boyle AJ, Chuang J, Farrar DJ, Starling RC. Accuracy of Seattle Heart Failure Model and HeartMate II Risk Score in Non-Inotrope-Dependent Advanced Heart Failure Patients: Insights From the ROADMAP Study (Risk Assessment and Comparative Effectiveness of Left Ventricular Assist Device and Medical Management in Ambulatory Heart Failure Patients). Circ Heart Fail. 2017 May;10(5):e003745. doi: 10.1161/CIRCHEARTFAILURE.116.003745. PMID 28465311
- [Derived] Starling RC, Estep JD, Horstmanshof DA, Milano CA, Stehlik J, Shah KB, Bruckner BA, Lee S, Long JW, Selzman CH, Kasirajan V, Haas DC, Boyle AJ, Chuang J, Farrar DJ, Rogers JG; ROADMAP Study Investigators. Risk Assessment and Comparative Effectiveness of Left Ventricular Assist Device and Medical Management in Ambulatory Heart Failure Patients: The ROADMAP Study 2-Year Results. JACC Heart Fail. 2017 Jul;5(7):518-527. doi: 10.1016/j.jchf.2017.02.016. Epub 2017 Apr 5. PMID 28396040
- [Derived] Estep JD, Starling RC, Horstmanshof DA, Milano CA, Selzman CH, Shah KB, Loebe M, Moazami N, Long JW, Stehlik J, Kasirajan V, Haas DC, O'Connell JB, Boyle AJ, Farrar DJ, Rogers JG; ROADMAP Study Investigators. Risk Assessment and Comparative Effectiveness of Left Ventricular Assist Device and Medical Management in Ambulatory Heart Failure Patients: Results From the ROADMAP Study. J Am Coll Cardiol. 2015 Oct 20;66(16):1747-1761. doi: 10.1016/j.jacc.2015.07.075. PMID 26483097